CLINICAL TRIAL: NCT06510309
Title: A Phase II Study Using Rituximab Plus Venetoclax in the Front Line Treatment of Marginal Zone Lymphoma
Brief Title: Rituximab Plus Venetoclax in Front Line Marginal Zone Lymphoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gottfried von Keudell, MD PhD (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor-Investigator, Gottfried von Keudell, MD PhD, Sponsor Investigator, Beth Israel Deaconess Medical Center
Organization: Beth Israel Deaconess Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-711
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Lymphoma; Marginal Zone Lymphoma; MZL
Keywords: Lymphoma; Marginal Zone Lymphoma; MZL
MeSH Terms: conditions — Lymphoma; Lymphoma, B-Cell, Marginal Zone | interventions — venetoclax; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rituximab + Venetoclax (Experimental): 33 participants will be enrolled and will complete study procedures as follows:
  * Baseline visit with screening assessments, scans, and tumor and bone marrow biopsies.
  * Induction Period:
    * CT/MRI scans at week 4.
    * Weeks 1 - 4: Predetermined dose of Rituximab 1x weekly.
    * Weeks 5 - 8: Predetermined dose of Venetoclax 1x daily.
  * Maintenance Period:
    * CT/MRI scan on weeks 12, 36, 60, 84, and then every 6 months after week 96.
    * Predetermined dose of Venetoclax 1x daily for up to week 96, then once every 6 months.
    * Predetermined dose of Rituximab 1x weekly at weeks 12, 24, 36, and 48.
  * End of Treatment Visit: CT/MRI scan, tumor biopsy, and bone marrow biopsy.
  * Follow up: In-clinic visit at 1 year after finishing study drugs.
  Interventions: Drug: Venetoclax; Drug: Rituximab

INTERVENTIONS:
Drug: Venetoclax — B-cell lymphoma inhibitor, tablets taken orally per protocol.
  Other Names: ABT-199; GDC-199
Drug: Rituximab — Anti-CD20 monoclonal antibody, 10mL or 50 mL single-use vials, via intravenous (into the vein) infusion per protocol.
  Other Names: Riabni; Ruxience; Truxima; Rituxan; ABP 798; IDEC-C2B8; PF-05280586

SUMMARY:
The purpose of this study is to see if the combination of rituximab and venetoclax is effective in treating participants with untreated Marginal Zone Lymphoma (MZL).

The names of the study drugs involved in this study are:

* Venetoclax (a type of inhibitor)
* Rituximab (a type of antibody)

DETAILED DESCRIPTION:
This is a phase II study of rituximab plus venetoclax in participants with MZL who have not had prior chemotherapy. The purpose of this study is to see if the combination of rituximab and venetoclax is effective in treating Marginal Zone Lymphoma.

The U.S. Food and Drug Administration (FDA) has not approved venetoclax for MZL but it has been approved for other uses.

The FDA has approved rituximab as a treatment option for MZL.

The research study procedures include screening for eligibility, study treatment visits, Computerized Tomography (CT) scans, Magnetic Resonance Imaging (MRI) scans, Positron Emission Tomography (PET) scans, blood tests, bone marrow and tumor biopsies, and electrocardiograms.

Participants will receive study treatment for up to 24 months and will be followed for 1 year after discontinuation of the study drugs.

It is expected that about 33 people will take part in this research study.

Abbvie, Inc. is funding this research study by providing venetoclax.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed Marginal Zone Lymphoma
* Patients must have measurable disease as defined by at least one lymph node ≥1.5 cm or spleen > 13 cm
* Patients with intestinal MALT lymphoma must have disease that is detectable by EGD or colonoscopy with biopsy
* Patients with gastric MALT lymphoma must be h. pylori negative. Patients who are h. pylori positive are allowed if they have failed a trial of h. pylori eradication
* Patients with gastric MALT lymphoma who are h. pylori negative or who relapsed/refractory disease after h. pylori eradication must be ineligible form have refused or failed gastric radiation therapy
* Age ≥18 years
* ECOG performance status ≤1
* Life expectancy of greater than 2 years
* Participants must meet the following organ and marrow function as defined below:

  * Hemoglobin ≥8.0 g/dL
  * absolute neutrophil count ≥1,000 cells/mcL (In the event of documented bone marrow involvement, ANC must be ≥1500 cells/mcL)
  * platelets ≥50,000 cells/mm3
  * total bilirubin < 1.5 x institutional upper limit of normal (ULN) (In patients with Gilberts disease or documented liver involvement, total bilirubin < 3 X ULN will be allowed)
  * AST(SGOT)/ALT(SGPT) < 3 × institutional ULN unless elevation is caused by liver involvement with MZL
  * Creatinine within institutional ULN OR creatinine clearance >60mL/min for patients with creatinine levels above institutional normal (by Cockcroft-Gault estimate or 12-24h creatinine clearance measurements)
* Ability to understand and the willingness to sign a written informed consent document
* Patient must be able to swallow pills
* HIV-positive patients on combination antiretroviral therapy are eligible if their HIV is under adequate control with an antiretroviral regimen that has been stable for > 4 weeks, as long as the CD4 count is >300. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Patients with Hepatitis B surface antibody serum positivity due to poor immunization, as well as those with Hepatitis B core antibody positivity with negative PCR on antiviral therapy will be eligible

Exclusion Criteria:

* Patients who had prior systemic therapy including rituximab
* Patients who have had prior radiation therapy, with the following exceptions:

  * Palliative radiotherapy (RT) is allowed, but must be completed at least 1 week prior to treatment on this study, and prior to any baseline imaging studies or biopsies. Patients must meet criteria for measurable/assessable disease as outlined above after completion of RT.
  * Prior RT for gastric MALT is allowed, but must be completed at least 1 week prior to treatment on this study, and prior to any baseline imaging studies or biopsies. Patients must meet criteria for measurable/assessable disease as outlined above after completion of RT.
* Prior treatment with ibrutinib or other BTK inhibitor
* Patients with h. pylori-associated gastric MALT or stage I/II MZL will be excluded unless they are deemed to be unfit for radiation therapy with curative intent.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with uncontrolled hepatitis B or C or HIV infection are ineligible defined as patients with positive serologies and a detectable viral load by PCR.
* Patients with Hep B core ab positivity are allowed provided Hep B PCR is undetectable
* Pregnant women or participants unwilling to adhere to institutional guidelines for highly effective contraception for 12 months after the last dose of rituximab are excluded from this study because of documented risks of rituximab on fetal immunologic development and unknown effects of venetoclax on embryonic development. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with venetoclax, breastfeeding should be discontinued.
* Received moderate or strong CYP3A inhibitors (such as fluconazole, ketoconazole, and clarithromycin) within 7 days prior to the first dose of venetoclax.
* Received moderate or strong CYP3A inducers (such as rifampin, carbamazepine, phenytoin, St. John's Wort) within 7 days prior to the first dose of venetoclax.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate (CRR) | Up to 24 months
  Complete Response (CR) rate is defined as the proportion of participants achieving CR during study treatment. CR is defined based on RECIL criteria.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 24 months
  ORR will be measured as the proportion of participants that achieve a PR or CR per RECIL criteria.
Partial Remission (PR) Rate | Up to 24 months
  Partial remission (PR) rate is defined as the proportion of participants achieving partial remission RECIL criteria.
Median Progression Free Survival (PFS) | Up to 24 months
  PFS based on Kaplan-Meier methodology will be measured from the time the participant initiates treatment until the first occurrence of documented progression of disease or death from any cause, censored for participants alive without progression.
Median Overall Survival (OS) | Up to 36 months
  OS based on Kaplan-Meier methodology will be measured from the time the participant initiates treatment until death from any cause, censored for participants alive.
Median Event Free Survival (EFS) | Up to 24 months
  EFS will be measured from the time the participant initiates treatment until documented off therapy for any reason, censored for participants who remain on therapy.
Duration of Response (DOR) | Up to 24 months
  DoR will be measured from the time of initial response until documented progression of disease, censored for participants who remain in response.

CONTACTS AND LOCATIONS:
Overall Officials: Gottfried von Keudell, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu